CLINICAL TRIAL: NCT05376631
Title: Effect of Fresh Gas Flow on Emergence Time in the Patients Undergoing Transurethral Resection of Bladder Tumor: A Randomized Controlled Clinical Trial
Brief Title: Effect of Fresh Gas Flow on Emergence Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, MD, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-0606
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Five (Active Comparator): For emergence from general anesthesia, a fresh gas flow of 5 L/min is used.
  Interventions: Procedure: Fresh gas flow of 5 L/min
- Group Ten (Experimental): For emergence from general anesthesia, a fresh gas flow of 10 L/min is used.
  Interventions: Procedure: Fresh gas flow of 10 L/min

INTERVENTIONS:
Procedure: Fresh gas flow of 5 L/min — A fresh gas flow of 5 L/min is used during emergence from general anesthesia.
  Arms: Group Five
Procedure: Fresh gas flow of 10 L/min — A fresh gas flow of 10 L/min is used during emergence from general anesthesia.
  Arms: Group Ten

SUMMARY:
The purpose of this study is to evaluate the effect of fresh gas flow on emergence time in patients undergoing transurethral resection of bladder tumor.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of fresh gas flow (5 L/min vs. 10 L/min) on emergence time in patients undergoing transurethral resection of bladder tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled transurethral resection of bladder tumor under general anesthesia
* Patients aged between 20 and 79 years old
* American Society of Anesthesiologists physical status ≤2
* Patients who are voluntarily agreed to this clinical study

Exclusion Criteria:

* A long operation (2 hours or longer)
* Hearing disturbance
* Cognitive disorder
* Psychiatric substance abuse
* Patient's denial

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Emergence time | From end of surgery to extubation (assessed up to 30 minutes after surgery)
  When consciousness and self respiration are fully recovered after surgery is ended, extubation is tried. The time to extubation (emergence time) is recorded.

SECONDARY OUTCOMES:
Time to spontaneous movement | From end of surgery to spontaneous movement (assessed up to 30 minutes after surgery)
  After surgery is stopped, the patients are asked to open their eyes every 1 minute after the termination of sevoflurane administration. The time to spontaneous movement is recorded.
Time to eye opening | From end of surgery to eye opening (assessed up to 30 minutes after surgery)
  After surgery is stopped, the patients are asked to open their eyes every 1 minute after the termination of sevoflurane administration. The time to eye opening is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaya da Costa M, Kalmar AF, Struys MMRF. Inhaled Anesthetics: Environmental Role, Occupational Risk, and Clinical Use. J Clin Med. 2021 Mar 22;10(6):1306. doi: 10.3390/jcm10061306. PMID 33810063
- [Background] Brioni JD, Varughese S, Ahmed R, Bein B. A clinical review of inhalation anesthesia with sevoflurane: from early research to emerging topics. J Anesth. 2017 Oct;31(5):764-778. doi: 10.1007/s00540-017-2375-6. Epub 2017 Jun 5. PMID 28585095
- [Background] Baum JA. Low-flow anesthesia: theory, practice, technical preconditions, advantages, and foreign gas accumulation. J Anesth. 1999;13(3):166-74. doi: 10.1007/s005400050050. No abstract available. PMID 14530937
- [Background] Sakata DJ, Gopalakrishnan NA, Orr JA, White JL, Westenskow DR. Hypercapnic hyperventilation shortens emergence time from isoflurane anesthesia. Anesth Analg. 2007 Mar;104(3):587-91. doi: 10.1213/01.ane.0000255074.96657.39. PMID 17312214
- [Background] Difficult Airway Society Extubation Guidelines Group; Popat M, Mitchell V, Dravid R, Patel A, Swampillai C, Higgs A. Difficult Airway Society Guidelines for the management of tracheal extubation. Anaesthesia. 2012 Mar;67(3):318-40. doi: 10.1111/j.1365-2044.2012.07075.x. PMID 22321104
- [Derived] Park JY, Yu J, Kim CS, Baek JW, Jo Y, Kim YK. Comparison of the effects of 5 and 10 L/minute fresh gas flow on emergence from sevoflurane anesthesia: A randomized clinical trial. Medicine (Baltimore). 2023 Jul 21;102(29):e34406. doi: 10.1097/MD.0000000000034406. PMID 37478213